CLINICAL TRIAL: NCT05192330
Title: The Effect of Virtual Reality Glasses Use and Therapeutic Touch on Pain, Anxiety and Patient Satisfaction in Women During Intrauterine Insemination Procedure: A Randomized Controlled Study
Brief Title: Intrauterine Insemination and Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/350
Record Dates: First submitted 2022-01-12; First posted 2022-01-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Infertility
Keywords: intrauterine insemination; nursing; pain; anxiety
MeSH Terms: conditions — Infertility; Pain; Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This randomized controlled study will conduct at Ondokuz Mayis University Training and Research Hospital, Obstetrics and Gynecology polyclinic between January 2022 and June 2022. The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomised controlled trials (RCTs) has been used to describe the methods.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (Experimental): After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and visual analogue scale(pain and nursing satisfaction) scoring scale will apply to both groups by face to face interview during the day giving appointment for intrauterine insemination. Immediately after the questionnaires were applied, the nurse gave Virtual Reality Glasses for 30 minutes.
  Glasses will be given put on before the process starts and training will be given to continue watching the video while wearing the glasses.The women include in the Virtual reality application group will be shown a video with a nature view during the procedure.
  Every woman will be shown the same video.
  Interventions: Device: Virtual Reality Glasses
- Therapeutic Touch (Experimental): Applied therapeutic touch intervention on their hands for 30 minutes to help patients feel comfortable during the procedure.The researcher started the application by taking an appropriate hand of the patient between his hands and held it for 30 minutes. The researcher's fingers are closed, not clasped, and his hand is placed on the participant's hand.
  The researcher held her hand steady without touching or rubbing it. In addition, the researcher is not use gloves.
  Interventions: Behavioral: Therapeutic Touch
- control group (No Intervention): Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (virtual reality or Therapeutic Touch) was performed. Both groups were re-evaluated using the same scales after the intrauterine insemination. Within 5 minutes of completing the procedure, participants will asked to evaluate their pain in order to characterize pain intensity using the visual analogue scale, anxiety scale and satisfaction scale.

INTERVENTIONS:
Device: Virtual Reality Glasses — After obtaining informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale (pain) were applied to both groups by face to face interview during the day giving appointment for intrauterine insemination. Immediately after the questionnaires were answered, virtual reality glasses were given by the nurse researcher to intervention group for 30 minutes.
  Arms: Virtual Reality Glasses
Behavioral: Therapeutic Touch — After obtaining informed consent, the data collection form, Spielberger State Anxiety Scale and VAS (pain) scoring scale were applied to both groups by face to face interview during the day giving appointment for intrauterine insemination. Immediately after the questionnaires were answered, therapeutictouch were given by the nurse researcher to intervention group for 30 minutes.
  Arms: Therapeutic Touch

SUMMARY:
This study investigates the effect of virtual reality glasses use and therapeutic touch on pain, anxiety and patient satisfaction in women during intrauterine insemination procedure

DETAILED DESCRIPTION:
Infertility treatment is a stressful and anxious process that begins when couples are diagnosed with infertility. Infertility treatment is a process that requires the active participation of couples against emotional and physical difficulties. In addition to intensive routine and surgical procedures, the treatment process is a period in which couples should be in constant communication with healthcare professionals. In Turkey, it is estimated that 10-20% of the couples are diagnosed with infertility. In the evaluation of infertile couples,Intrauterine Insemination is a simple, safe, and minimally invasive procedure to the process of injecting washed sperm into the uterine cavity close to ovulation. Sperm cells taken from men are injected directly into the uterus and left at a point closer to the fertilization point. The aim of this study is to investigate the effect of virtual reality glasses use and therapeutic touch on pain, anxiety and patient satisfaction in women during intrauterine insemination procedure.

This randomized controlled study will conduct at Ondokuz Mayis University Training and Research Hospital, Infertility polyclinic between january 2022 and June 2022.

Volunteer women undergoing Intrauterine Insemination will be include. Participants will randomly assigned to the intervention or the control group using a computer-generated list. A data collection form including socio-demographic and obstetric characteristics such as age, educational status, duration of infertility, previous pregnancies, births, abortion/curettage numbers, Spielberger State Anxiety Scale and Visual Analog Scale scores will use for each patient. After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale (pain and nursing satisfaction) were applied to both groups by face to face interview during the day giving appointment for Intrauterine Insemination. Immediately after the questionnaires will apply, the nurse gave virtual reality glasses. and glasses will be put on before the process starts and training will be given to continue watching the video while wearing the glasses for 30 minutes. Second group participants the nurse researcher will start the application by taking an appropriate hand of the patient between his hands and hold it for 30 minutes.

Participant in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (virtual reality or therapeutic touch) was performed.The IBM SPSS (Statistical package for the Social Sciences) 23.0 package program was used to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

being diagnosed with infertility over 18 years, being able to understand, read and write in Turkish, wanting to participate in the study,

Exclusion Criteria:

not wanting to be included in the study not accepting Therapeutic Touch or Virtual reality glasses not knowing Turkish not wanting to be included in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Spielberger State Anxiety Scale | 30 minutes
  After completing the Intrauterine Insemination Procedure, participants filled out the Spielberger State Anxiety Scale.
  The inventory was developed by Spielberger, Gorsuch, and Lushene in 1970. An adaptation, validity, and reliability study of the State-Trait Anxiety Scale in Turkish was conducted by Oner and Le Compte in 1983. The scale consists of two subdimensions: the state anxiety has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the trait anxiety has 20 items and is used to determine what has been felt in the last 7 days. High scores from each subscale indicate a high level of anxiety.
Visual Analog Scale for pain intensity | 10 minutes
  After completing the Intrauterine Insemination Procedure, participants were asked to evaluate their pain in order to characterize pain intensity using the Visual Analog Scale (VAS).
  A standard ten-point visual analogue scale (VAS) of 0 to 10 was designed and used to assess the patients' perceptions of discomfort during the procedure. A high score on the scale indicated a high level of discomfort and a score of 0 denoted no discomfort at all. Patients indicate the degree of pain they feel between 0-10.
Visual Analog Scale for patient satifaction | 10 minutess
  Satisfaction level was measured using the visual analog scale (VAS). VAS is used to convert some numerically unmeasured values to numeric values. VAS is a continuous scale that comprises a horizontal line or a vertical line, usually 10 cm (100 mm) in length. On one end of the scale is the statement, "I am not satisfied at all" (zero points), whereas the statement at the other end is "very satisfied." Patients were asked to mark their satisfaction levels on this scale of 100 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Emine KOÇ, Asst.Prof, Study Chair — Ondokuz Mayıs University; Neşe KARAKAYA, lecturer, Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Nazarinasab, M., Motamedfar, A., Najafian, M., & Tabibi, H. (2018). Investigating the effects of relaxation therapy on decreasing anxiety in patients with elective caesarean section in Imam Khomeini Hospital, Ahvaz, Iran during 2016. Medical Studies/Studia Medyczne, 34(2), 107-111.
- [Derived] Bal S, Karakaya N, Koc E, Guven D. The effect of virtual reality (VR) glasses and therapeutic touch (TT) on pain, anxiety, and patient satisfaction during intrauterine insemination (IUI) compared to standard care: a single-blind, randomized controlled trial. BMC Pregnancy Childbirth. 2025 Mar 27;25(1):361. doi: 10.1186/s12884-025-07435-0. PMID 40148795